CLINICAL TRIAL: NCT06075394
Title: The Effect of Antihypertensive Medication Usage on the Status of Psoriasis in Patients Concurrently Having Hypertension.
Brief Title: Hypertension, Antihypertensive Medication Use, and Risk of Psoriasis
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, chief of dermatology, Xijing Hospital
Other Study IDs: xijingH-PF-202310
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Psoriasis
Keywords: Hypertension; Antihypertensive Medication; Psoriasis
MeSH Terms: conditions — Psoriasis; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psoriasis patients: Patients with psoriasis in the Department of Dermatology, Xijing Hospital of Air Force Medical University from December 2012 to December 2022 were consecutively collected. Inclusion criteria: (1) age ≥18 years; (2) Clear diagnosis of psoriasis. Exclusion criteria: (1) age <18; (2) Hypertension caused by conditions such as primary hypertension, hyperthyroidism, chronic renal insufficiency, or Cushing's syndrome, which are severe endocrine system diseases; (3) Patients with autoimmune diseases, severe cardiovascular, hepatic, renal, or other major organ disorders, as well as blood disorders and endocrine system diseases.
- Healthy individuals: Healthy individuals being randomly selected healthy individuals from a medical examination center.

SUMMARY:
The influences of hypertension and antihypertensive medication on psoriasis have been long discussed. Given the limited and inconsistent evidence available, there is a need to further explore and clarify the relationship between hypertension and psoriasis, as well as to assess the relationship between antihypertensive medication use and the development or worsening of psoriasis symptoms. The aim of this retrospective study was to analyze data from electronic health records in a large population-based cohort, and the investigators aimed to investigate whether there was a significant association between hypertension and the use of related antihypertensive medications, such as ACEis, and psoriasis, and to explore potential confounders that may influence this association. Understanding the potential relationship between antihypertensive medication and psoriasis is critical, as this may have implications for the management of hypertension in patients with psoriasis or those at risk of developing the condition. This study will contribute to the existing body of evidence and provide valuable insights for clinicians to make informed decisions about the use of antihypertensive medication in this patient population, ultimately contributing to more effective prevention and management strategies for individuals affected by these diseases.

DETAILED DESCRIPTION:
The investigators conducted a retrospective cohort study of psoriasis patients (≥18 years old) admitted as inpatients of Xijing hospital. Prior to the commencement of the survey, the investigators underwent collective training on data collection procedures to ensure the quality and reliability of the data. The study population included psoriasis patients aged 18 years or older who had been hospitalized at least once between 2012 and December 2022. Healthy individuals being randomly selected healthy individuals from a medical examination center. According to local ethics, the investigators have applied for exemption from written informed consent.

Patients with psoriasis in the Department of Dermatology, Xijing Hospital of Air Force Medical University from December 2012 to December 2022 were consecutively collected. Inclusion criteria: (1) age ≥18 years; (2) Clear diagnosis of psoriasis. Exclusion criteria: (1) age <18; (2) Hypertension caused by conditions such as primary hypertension, hyperthyroidism, chronic renal insufficiency, or Cushing's syndrome, which are severe endocrine system diseases; (3) Patients with autoimmune diseases, severe cardiovascular, hepatic, renal, or other major organ disorders, as well as blood disorders and endocrine system diseases.

The study collected various parameters, including baseline information such as ID number, gender, date of birth, medical history, and family history. Psoriasis-related data included age at first onset, date of diagnosis, duration of disease, frequency of relapse, psoriasis subtype, history of systemic/local medication, and comorbidities such as hypertension and dyslipidemia.

Furthermore, clinical examination data and laboratory tests were conducted, which included measurements such as height, weight, systolic blood pressure (SBP), diastolic blood pressure (DBP), PASI score (Psoriasis Area and Severity Index), fasting plasma glucose (FPG), total cholesterol (TC), total triglycerides, uric acid, neutrophil count (normal range 1.80-6.30 × 109/L), and lymphocyte count (normal range 1.00-4.80 × 109/L). It is important to note that all blood tests were conducted prior to any treatment.

The above information was obtained from the Medical Record System of Xijing Hospital of Air Force Medical University.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Clear diagnosis of psoriasis

Exclusion Criteria:

* Age <18;
* Hypertension caused by conditions such as primary hypertension, hyperthyroidism, chronic renal insufficiency, or Cushing's syndrome, which are severe endocrine system diseases;
* Patients with autoimmune diseases, severe cardiovascular, hepatic, renal, or other major organ disorders, as well as blood disorders and endocrine system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators conducted a retrospective cohort study of psoriasis patients (≥18 years old) admitted as inpatients of Xijing hospital. Prior to the commencement of the survey, the investigators underwent collective training on data collection procedures to ensure the quality and reliability of the data. The study population included psoriasis patients aged 18 years or older who had been hospitalized at least once between 2012 and December 2022. Healthy individuals being randomly selected healthy individuals from a medical examination center.
Sampling Method: Non-Probability Sample
Enrollment: 9294 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Hypertension as a risk factor for psoriasis | Information collection: over a span of 2 months
  Hypertension has the potential to act as an underlying risk factor for the onset of psoriasis and has been identified as correlating with the frequency of recurrent psoriatic episodes.

SECONDARY OUTCOMES:
Antihypertensive Medication as a risk factor for psoriasis | Information collection: over a span of 2 months
  The use of antihypertensive medication may serve as a contributing factor to the risk of psoriatic relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China